CLINICAL TRIAL: NCT02995681
Title: Randomized Controlled Trial of Balance Training for Fall Reduction in Individuals With COPD
Brief Title: Balance Training for Fall Reduction in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic restrictions
Sponsor: West Park Healthcare Centre (Other)
Collaborators: University of British Columbia (Other); Dalhousie University (Other); University of Alberta (Other); University of Ottawa (Other); Teesside University (Other); University of Sydney (Other); La Trobe University (Other); Aveiro University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Respirologist, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-018-WP
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Copd; Fall Patients
Keywords: COPD; Falls; Balance training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary rehab and balance training (Experimental): The intervention group will receive standard pulmonary rehab plus additional balance training.
  Interventions: Other: Balance training; Other: Pulmonary rehab
- Pulmonary rehab (Active Comparator): The control group will receive pulmonary rehab only and a pulmonary rehab home program (walking and lower extremity resistance exercises) upon discharge from pulmonary. They will also receive the same monthly phone calls and three home visits at three, six and nine months to ensure proper technique and progression.
  Interventions: Other: Pulmonary rehab

INTERVENTIONS:
Other: Balance training — Balance exercises will include: functional lower extremity training, gait training under challenging conditions and training to increase stability during changes in body positions.
  Arms: Pulmonary rehab and balance training
Other: Pulmonary rehab — Pulmonary rehab includes: supervised exercise (aerobic exercise, resistance exercise) disease-specific education, and psychological and social support.

SUMMARY:
People living with Chronic Obstructive Pulmonary Disease (COPD) have problems with their balance and a high incidence of falls compared to those of a similar age. Pulmonary rehabilitation is recommended for people with COPD, however, these training programs do not typically include balance training or fall prevention strategies. In this study, patients with COPD who report problems with their balance or have had a fall in the last two years will be assigned to a treatment group (balance training plus pulmonary rehabilitation) or control group (standard pulmonary rehabilitation). We will record the number of falls using monthly diaries and evaluate patient's balance, strength, confidence and quality of life.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality in Canada. In addition to lung impairment, secondary effects of the disease are well established including impairments in muscle function and exercise capacity. However, individuals with COPD also have marked deficits in balance and an increased risk of falls with a 3-5 times higher annual fall rate than those of similar age. The underlying mechanisms remain unclear, but several factors have been implicated including decreased physical activity, muscle weakness, altered trunk mechanics, comorbidities, hypoxemia and proprioceptive deficits. Given this unique impairment profile, tailored approaches to balance training and fall prevention are needed in COPD.

Pulmonary rehabilitation (PR) is an integral therapeutic intervention for individuals with COPD. The program typically consists of supervised exercise, disease-specific education, and psychological and social support. Balance training and fall prevention strategies are not currently included in international guidelines for PR and few programs include any balance assessment. We have previously shown that the exercise component of traditional PR has minimal effect on measures of balance and fall risk. We then conducted an RCT to examine the effects of balance training alongside PR, which specifically addressed the profile of balance deficits we had identified in COPD. Tailored balance training alongside PR results in clinically important improvements in balance performance compared to PR alone. Given these results, we now have the opportunity to build on our existing experience to test the effect of the intervention on falls.

The purpose of this study is to establish the efficacy of a tailored balance exercise program for reducing falls in individuals with COPD enrolled in PR. If participation in tailored balance training decreases falls compared to usual PR, this approach will represent an innovative and potential cost-saving strategy to prevent falls and reduce associated healthcare utilization in COPD. Our results will be relevant for guiding clinical and policy-based decision making, given the large population of individuals with COPD and the potential for severe consequences of falls in this population.

The primary objective of this study is to evaluate the long-term effects of tailored balance exercise on the rate of falls in individuals with COPD enrolled in PR. Secondary objectives are to determine 1) the long-term effects of the program on measures of balance, balance confidence and muscle strength; and 2) the cost-utility of the program.

ELIGIBILITY:
Inclusion Criteria:

* a physician diagnosis of COPD based on GOLD criteria; a self-reported decline in balance, a fall within the last two years or a recent near fall; and an ability to provide written informed consent

Exclusion Criteria:

* severe cognitive impairment (dementia, neurological condition) an inability to communicate because of language skills (aphasia, non-English speaking), or evidence of a neurological or musculoskeletal condition that severely limits mobility and postural control (e.g. cerebrovascular accident, Parkinson's Disease, amputation) and may jeopardize their safety or influence their balance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-01; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Number of falls | 12 months
  Number of falls will be measured using monthly falls diaries

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Clinical measure of balance
Balance Evaluation Systems Test (BESTest) | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Clinical measure of balance
Activities Specific Balance Confidence Scale | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Balance confidence questionnaire
30 Second Repeated Chair Stand Test | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Functional lower body strength test
European Quality of Life 5-Dimension Questionnaire (EQ-5D-5L) | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 6 months, 12 months
  Health status questionnaire

OTHER OUTCOMES:
Baseline Dyspnea Index | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Descriptive measure of shortness of breath
Falls Risk for Older People - Community Setting (FROP-Com) | Baseline (pre pulmonary rehab), 8 weeks (post pulmonary rehab), 12 months
  Descriptive measure of falls risk in community dwelling older people

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — West Park Healthcare Centre; Roger Goldstein, MD, Principal Investigator — West Park Healthcare Centre; Marla Beauchamp, PhD, Principal Investigator — West Park Healthcare Centre
Locations (10):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Alfred Health, Melbourne, Victoria
  - Western Health, Saint Albans, Victoria
- Canada (5):
  - G.F. Macdonald Centre for Lung Health, Edmonton, Alberta
  - St. Paul's Pulmonary Rehab Program, Vancouver, British Columbia
  - Colchester East Hants Health Authority, Truro, Nova Scotia
  - Ottawa Hospital Rehabilitation Centre, Ottawa, Ontario
  - West Park Healthcare Centre, Toronto, Ontario
- School of Health Sciences, University of Aveiro, Aveiro, Portugal
- James Cook University Hospital, Middlesbrough, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen KT, Brooks D, Macedo LG, Ellerton C, Goldstein RS, Alison J, Dechman G, Harrison S, Holland AE, Lee A, Marques A, Spencer L, Stickland MK, Skinner EH, Haines KJ, Beauchamp MK. Development of a clinical prediction model for falls in individuals with COPD. BMJ Open Respir Res. 2025 Dec 25;12(1):e002556. doi: 10.1136/bmjresp-2024-002556. PMID 41448796
- [Derived] Hao Q, Brooks D, Ellerton C, Goldstein R, Lee AL, Alison JA, Dechman G, Haines KJ, Harrison SL, Holland AE, Marques A, Spencer L, Stickland MK, Skinner EH, Camp PG, Ma J, Beauchamp MK. Pulmonary rehabilitation with balance training for fall reduction in chronic obstructive pulmonary disease: a randomized controlled trial. BMC Pulm Med. 2024 Aug 24;24(1):408. doi: 10.1186/s12890-024-03215-2. PMID 39182033
- [Derived] Beauchamp MK, Brooks D, Ellerton C, Lee A, Alison J, Camp PG, Dechman G, Haines K, Harrison SL, Holland AE, Marques A, Moineddin R, Skinner EH, Spencer L, Stickland MK, Xie F, Goldstein RS. Pulmonary Rehabilitation With Balance Training for Fall Reduction in Chronic Obstructive Pulmonary Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Nov 20;6(11):e228. doi: 10.2196/resprot.8178. PMID 29158206